CLINICAL TRIAL: NCT02569333
Title: Patient Centered Algorithms to Optimize the Inpatient Experience and Treatment of Ulcerative Colitis: PATIENT-UC
Brief Title: Patient Centered Algorithms to Optimize the Inpatient Experience and Treatment of Ulcerative Colitis
Acronym: PATIENT-UC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of British Columbia (Other); University of Calgary (Other); University of Manitoba (Other); University of Ottawa (Other); McGill University (Other); University of Alberta (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Abbvie-PATIENT-UC
Record Dates: First submitted 2015-09-29; First posted 2015-10-06 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases; Colitis; Intestinal Disease
Keywords: ulcerative colitis; inflammatory bowel disease; education; patient-reported outcomes
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Colitis; Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Video (Experimental): Subjects to have access to educational video during hospital stay
  Interventions: Other: Educational video
- Usual Care (No Intervention): Patients to receive usual care and will not have access to educational video.

INTERVENTIONS:
Other: Educational video — iPad with educational video highlighting current guidelines for the management of hospitalized patients with ulcerative colitis.
  Arms: Educational Video

SUMMARY:
Hospitalized patients with ulcerative colitis (UC) are at increased risk for a variety of complications such as infections, venous thrombosis, and surgery. The literature has revealed significant variation in the quality of care to hospitalized UC patients. As a result, guidelines for the management of these patients have been developed. However, the update of guidelines are variable. Admission to hospital can also have significant impact on quality of life due to interruptions in life commitments and lost sense of control of disease. Maintaining a sense of self-control of disease and active participation in care has been shown to be valuable among individuals with chronic diseases. The investigators propose the development of a multi-site, patient centred initiative aimed at improving clinical and patient-centered outcomes through an educational iPad based tool for patients admitted to hospital with ulcerative colitis.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic gastrointestinal condition with significant morbidity in the form of hospitalizations, surgery, and reductions in quality of life. Most patients with IBD are managed in an ambulatory, outpatient setting. However, to optimally manage severe disease activity, hospitalization may be required. Hospitalized patients are at increased risk for a variety of complications such as infections, venous thrombosis, and surgery. The literature has revealed significant variation in care and disease outcomes among hospitalized IBD patients. The heterogeneous nature of IBD severity, location, and phenotype as well as limited evidence to guide some therapeutic domains make standardization of IBD care delivery difficult. However, hospitalized patients with ulcerative colitis (UC) represent a more homogenous group that may be most amendable to quality improvement initiatives aimed at reducing variation, a known surrogate marker of poor performance. The Canadian Association of Gastroenterology has developed guidelines for hospitalized UC patients. It is well established, however, that update of guidelines are variable.

Admission to hospital can also have significant impact on quality of life due to interruptions in life commitments and lost sense of control of disease. Maintaining a sense of self-control of disease and active participation in care has been shown to be valuable among individuals with chronic diseases such as IBD. The investigators proposed the development of a multi-site, patient centered initiative aimed at improving clinically relevant and patient-centered outcomes through a multi-faceted educational tool for patients admitted to hospital with ulcerative colitis. Participating sites will be randomized to usual care versus administering the educational tool to patients which outlines what to expect during their hospital stay and reviews the current guidelines for hospitalized ulcerative colitis management.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ulcerative colitis
* able to provide informed consent
* admission to hospital with flare of underlying ulcerative colitis

Exclusion Criteria:

* Crohn's disease
* inability to provide informed consent
* readmission during study period (intervention would only be used on the initial admission during the study period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Overall length of stay | 1 year
Percentage of patients undergoing colectomy | 1 year

OTHER OUTCOMES:
Proportion of patient undergoing testing of C difficile within 48 hours of admission | 1 year
Time from initiation of IV steroids to salvage therapy or surgery. | 1 year
Proportion of patients receiving VTE prophylaxis | 1 year
Trust in physician as measured by TIPS | 6 months
Patient Satisfaction as measured by CACHE | 6 months
Anxiety and Depression as measured by HADS. | 6 months
Adherence to Medication as measured by Morisky scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam V. Weizman, MD, MSc, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Weizman AV, Bressler B, Seow CH, Afif W, Afzal NM, Targownik L, Nguyen DM, Jones JL, Huang V, Murthy SK, Nguyen GC. Providing Hospitalized Ulcerative Colitis Patients With Practice Guidelines Improves Patient-Reported Outcomes. J Can Assoc Gastroenterol. 2020 Jun 9;4(3):131-136. doi: 10.1093/jcag/gwaa019. eCollection 2021 Jun. PMID 34061122